CLINICAL TRIAL: NCT01020318
Title: Evaluation of Outcome Measures for Patients Diagnosed With Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: United States Department of Defense (U.S. Federal Agency); Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Other Study IDs: 100006; 10-CC-0006
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2014-05-16

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; TBI; Brain Injuries
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Traumatic brain injury (TBI) is a significant injury in the Armed Forces, but it is also common in the general population. This condition poses significant challenges for both diagnosis and therapy. However, the biological and neurological reasons for TBI remain poorly understood and are in need of more in-depth study.
* The National Institutes of Health is collaborating with several military medical centers and research units in a multi-year study of TBI in civilian and military patients. In anticipation of these research projects, the Clinical Center s Rehabilitation Medicine Department needs to become familiar with the instruments they will likely need to evaluate this group of subjects.

Objectives:

* To evaluate potential test instruments in patients with TBI.
* To evaluate patient tolerance of an extensive battery of assessments and the time required to complete the assessments.
* To improve staff competencies on new or novel assessments of the TBI patient population

Eligibility:

* Individuals 18 years of age and older who have been diagnosed with a traumatic brain injury in the past 5 years.
* Healthy volunteers 18 years of age and older who have had no instances of significant head trauma.

Design:

* This study requires approximately 3 days of outpatient or inpatient evaluation.
* Subjects will undergo cognitive and neuropsychological tests, physical assessments, speech and language evaluation, and balance testing. Tests will be given orally, in writing, and on computers. The testing will be done in blocks of 2 to 3 hours, with rest periods as needed.
* Subjects may undergo any or all of the following assessments and screening tools, as determined by the researchers:
* Cognitive, quality of life, and functional assessments
* Speech, language, and swallowing assessments
* Physical functional performance and environment assessments (including balance testing)
* Subjects will remain under the care of their own health care providers while participating in this study.

DETAILED DESCRIPTION:
The objective of this study is to evaluate potential test instruments in the traumatic brain injury (TBI) patient population. We will assess outcome measures that test neuropsychological, cognitive, communicative, and physical functional outcomes on up to 60 patients with TBI and 20 healthy volunteers. Our aims are to evaluate the appropriateness of specific tests for TBI as well as to test patient tolerance of an extensive battery of assessments and the time required to complete the assessments. We will also focus on improving staff competencies as they relate to new or novel assessments on the TBI patient population.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. For TBI patients: a diagnosis of TBI within the last 5 years
  2. For Healthy volunteers: no episode of head trauma resulting in an alteration in level of consciousness or loss of memory for the event.

EXCLUSION CRITERIA:

For both study populations:

1. Age less than 18 years
2. Inability to speak or understand English well enough to complete study instruments
3. Medically unstable on evaluation by an RMD physician, including those with clinically significant medical conditions that would make the research evaluations unsafe, logistically difficult or impossible to complete.
4. Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-10-16; Study Completion 2014-05-16

CONTACTS AND LOCATIONS:
Overall Officials: Leighton Chan, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States